CLINICAL TRIAL: NCT01955174
Title: Endoscopic Injection of Botulinum Toxin in Patients With Hypercontractile Esophageal Motility Disorders: a Prospective, Randomized, Double-blind, Controlled Study
Brief Title: Botulinum Toxin Injection in Hypercontractile Esophagus
Acronym: TIBOH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012.779
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Nutcracker Oesophagus
Keywords: Botulinum toxin; Esophageal motility disorder; Distal esophageal spasm
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin injection (Experimental): Esophageal endoscopic injection of botulinum toxin
  Interventions: Drug: Esophageal endoscopic injection of botulinum toxin
- No injection (Sham Comparator): No injection of botulinum toxin
  Interventions: Other: No injection of botulinum toxin

INTERVENTIONS:
Drug: Esophageal endoscopic injection of botulinum toxin — Endoscopic injection of botulinum toxin in the esophageal muscle : one hundred units of type A botulinum toxin (Botox®, Allergan) diluted in 10 mL of normal saline and injected at the lower third of the esophageal wall in 10 sites between 2 and 10 cm above the Z-line.
  Arms: Botulinum toxin injection
Other: No injection of botulinum toxin — Upper gastro-intestinal endoscopy without any injection
  Arms: No injection

SUMMARY:
This study aims to evaluate the efficacy and the safety of endoscopic injection of 100 IU of botulinum toxin (BTX) in the distal esophagus in patients with symptoms related to hypercontractile esophageal motility disorders.

DETAILED DESCRIPTION:
Eligible patients will present chest pain and/or dysphagia related to the following hypercontractile esophageal motility disorders: distal esophageal spasm, jackhammer esophagus, nutcracker esophagus or type III achalasia with normalization of the integrated relaxation pressure after treatment, based on the Chicago classification of esophageal motility disorders for high resolution manometry (HRM). Upper gastrointestinal endoscopy and barium swallow will be performed before BTX injection to eliminate secondary disorders.

This is a prospective, randomized, double blind, controlled trial comparing BTX injection to sham procedure (absence of injection, the clinical team performing the follow-up will not be aware of the result of the randomization).

Drugs which could affect esophageal motility (nitrates and calcium channel blockers) will be stopped during the study.

Included patients will undergo esophageal endoscopic ultrasound examination (EEUS) and upper gastrointestinal endoscopy under general anesthesia. In absence of contraindications, patients will be randomized in two arms: BTX injection or no injection. The active treatment group will receive 100 units of type A BTX (Botox®, Allergan) diluted in 10 mL of saline serum; BTX will be injected into the lower third of the esophageal wall in 10 sites between 2 and 10 cm above the squamo-columnar junction. The control arm will receive no injection after the EEUS and upper GI endoscopy (sham procedure).

Clinical response will be assessed based on the evolution of the Eckardt score, a quality of life score (Gastrointestinal Quality of Life Index (GIQLI), and weight gain. A significant clinical response will be defined as an Eckardt score < 3 (together with individual scores < 2). Manometry patterns will be compared before and after the procedure. Safety will be monitored based on the occurrence of chest pain scored on a Likert scale and occurrence of adverse events.

Follow-up clinical evaluation will be performed 1 and 2 months after the procedure. A second esophageal HRM will be realized 3 months after the procedure, followed by endoscopic BTX injection in case of non-response and two monthly visits.

Follow-up visits will be done 6 and 12 months after the first procedure. An additional HRM will be performed at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-cardiac chest pain and/or dysphagia with global Eckardt score strictly above 3 points or equal to 3 only for " chest pain " or " dysphagia " - Hypercontractile esophagus with normal esogastric junction relaxation based on the Chicago classification in high resolution manometry
* Man or woman 18-year old or older
* Normal upper gastrointestinal endoscopy within one year before inclusion
* Barium swallow without argument for external compression
* Effective form of birth control (if applicable)
* Signed written informed consent form voluntarily
* Patient with health insurance

Exclusion Criteria:

* Man or woman under 18-year old
* Past history of eso-gastric surgery
* Evolutive cancer or coagulation disorders
* Absence of effective form of birth control (if applicable)
* Pregnant woman or woman who plans to become pregnant during the expected length of the study
* Breastfeeding woman
* Allergy to botulinum toxin or excipients
* Myasthenia
* Aminoglycoside treatment
* Endoscopic contraindication prior to the study
* Endoscopic contraindication during the study
* Psychiatric or addictive disease which could affect compliance to the constraints of the study
* Patient refusing to participate to the study
* Language barrier limiting the understanding of the study
* Incapability to give consent
* Concomitant participation to another research study
* No written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Clinical response | 3 months after Botulinum toxin injection or sham procedure
  Determination of the percentage of patients with clinical response defined by a global Eckardt score <3 and individual subscores <2

SECONDARY OUTCOMES:
Clinical symptoms improvement | 12 months after Botulinum toxin injection or sham procedure
  Determination of the percentage of patients with clinical response defined by a global Eckardt score <3 and individual subscores <2
Clinical symptoms improvement | After 2 procedures of Botulinum toxin injection or sham procedure
  Determination of the percentage of patients with clinical response defined by a global Eckardt score <3 and individual subscores <2
Safety | Days 1- 7 after procedure. Month 1,3, 4, 6 and 12 after procedure
  Evaluation of chest pain with numerical scale from 0 (no pain) to 10 (worst pain) along the 15 days following the procedure, and percentage of patients experimenting adverse events.
Quality of life improvement | At the first visit, 3 months, 6 months and 12 months after the first therapeutic procedure (botulinum toxin injection or sham procedure)
  Evaluation of the quality of life with the Gastrointestinal Quality of Life Index (GIQLI)
Weight gain | 3 months, 6 months and 12 months after the first therapeutic procedure (botulinum toxin injection or sham procedure)
  Evaluation of weight in kg
Modification of HRM pattern | 3 and 12 months after the first procedure (botulinum toxin injection or sham procedure)
  Change towards normal of specific HRM metrics: decrease of mean Distal Contratile Integral, disappearance of contraction with DCI > 8 000, increase of the % of contractions with normal Distal Latency
Clinical and paraclinical characteristics of responders versus non-responders | 12 months after the first therapeutic procedure (botulinum toxin injection or sham procedure)
  Age, sex, BMI, associated diseases, esophageal motility disorder according to the Chicago classification, associated medications, severity of symptoms at baseline (Eckardt) score, impairment of QOL at baseline (GIQLI score)

CONTACTS AND LOCATIONS:
Overall Officials: François MION, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service d'Hépato-Gastro-Entérologie et Oncologie Digestive- Hôpital Haut Lévêque - CHU de Bordeaux, Bordeaux
  - Service d'Exploration Fonctionnelle Digestive - Hôpital Edouard Herriot Pavillon H 5 - Hospices Civils de Lyon, Lyon

REFERENCES:
- [Result] Mion F, Marjoux S, Subtil F, Pioche M, Rivory J, Roman S, Zerbib F. Botulinum toxin for the treatment of hypercontractile esophagus: Results of a double-blind randomized sham-controlled study. Neurogastroenterol Motil. 2019 May;31(5):e13587. doi: 10.1111/nmo.13587. Epub 2019 Apr 11. PMID 30974039